CLINICAL TRIAL: NCT00533117
Title: Treating Suicidal Behavior and Self-Mutilation in Borderline Personality Disorder
Brief Title: Treating Suicidal Behavior and Self-Mutilation in People With Borderline Personality Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Beth Brodsky, Associate Director, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #5401R; R01MH061017-02 (NIH)
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Borderline Personality Disorder
Keywords: suicide; self-mutilation; fluoxetine; placebo; dialectical behavior therapy; supportive therapy
MeSH Terms: conditions — Borderline Personality Disorder; Suicide; Self-Injurious Behavior | interventions — Fluoxetine; Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dialectical Behavior Therapy Fluoxetine (Experimental): Dialectal behavior therapy (DBT) is a form of Cognitive behavior therapy (CBT) targeting suicidal and non-suicidal self injury in borderline personality disorder and is delivered over a 12 month period,and fluoxetine, a selective serotonin reuptake inhibitor (SSRI) that is given in standard dosing 20, 40, 60, 80 mg for 12 months.
  Interventions: Drug: Fluoxetine; Behavioral: Dialectical Behavior Therapy
- Dialectical Behavior Therapy placebo (Placebo Comparator): Dialectal behavior therapy and placebo Dialectal behavior therapy (DBT) is a form of Cognitive behavior therapy targeting suicidal and non-suicidal self injury in borderline personality disorder and is delivered over a 12 month period, and placebo for fluoxetine, an SSRI that is given in standard dosing 20, 40, 60, 80 mg for 12 months.
  Interventions: Behavioral: Dialectical Behavior Therapy
- Supportive therapy Fluoxetine (Experimental): Supportive psychotherapy and fluoxetine Supportive therapy is a manualized psychotherapy aimed at strengthening coping skills and is delivered over a 12 month period, and fluoxetine, an SSRI that is given in standard dosing 20, 40, 60, 80 mg for 12 months.
  Interventions: Drug: Fluoxetine; Behavioral: Supportive psychotherapy
- Supportive therapy placebo (Active Comparator): Supportive psychotherapy and placebo See above for descriptions.
  Interventions: Behavioral: Supportive psychotherapy

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine is administered in standard dosing 20, 40, 60, 80 mg increased monthly if tolerated
  Other Names: Prozac
  Arms: Dialectical Behavior Therapy Fluoxetine; Supportive therapy Fluoxetine
Behavioral: Dialectical Behavior Therapy — Dialectical Behavior Therapy is a form of CBT originally developed to treat suicidal and self injuring individuals with borderline personality disorder. Treatment consists of 2 sessions/week: individual psychotherapy and skills training group.
  Other Names: DBT
  Arms: Dialectical Behavior Therapy Fluoxetine; Dialectical Behavior Therapy placebo
Behavioral: Supportive psychotherapy — Supportive therapy is a manualized form of psychotherapy designed to enhance individual's strengths and coping mechanisms while reducing distress.
  Arms: Supportive therapy Fluoxetine; Supportive therapy placebo

SUMMARY:
This study will determine whether dialectical behavior therapy and fluoxetine are more effective combined or alone in treating people with borderline personality disorder.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) can be a serious and very complex condition. BPD affects 2% to 3% of the population and is more commonly diagnosed in young women. BPD is characterized by mood swings, impulsive behavior, difficulty controlling emotions, and acting out inappropriately either through self-harm or attempts of suicide. Other illnesses such as depression and anxiety are also very common in people diagnosed with BPD. Various treatments exist that aim to reduce self-harm and suicide among people with BPD. Dialectical behavior therapy (DBT), an outpatient behavioral therapy shown to help self-injurious patients with BPD, has become a popular treatment. Another useful treatment, the antidepressant fluoxetine, can help to regulate mood and diminish suicidal or self-destructive urges. Although combination treatments of DBT and fluoxetine are common, little research has been conducted on the effectiveness of this kind of combined treatment. The purpose of this study is to determine whether DBT and fluoxetine are more effective combined or alone in treating people with BPD.

All participants in this double-blind study will receive a psychiatric and medication evaluation prior to starting treatment. Participants taking psychiatric medications prior to the study will be slowly withdrawn from the medications over a period of 2 to 6 weeks. Psychological interviews and self-report questionnaires will be administered, taking approximately 5 to 10 hours to complete. Once all preliminary interviews and evaluations have been completed, each participant will be randomly assigned to one of the four following treatment groups:

* Group 1 will receive DBT and fluoxetine (Prozac). DBT teaches patients new skills to replace old coping strategies such as suicide attempts and self-injury. Participants will work with an individual therapist for 1 hour a week to learn these new skills. This group will also be expected to keep a weekly diary that will discuss their current mood; suicidal and self-harming urges; and possible use of medications, drugs, and alcohol. Once a week participants will engage in a 90-minute skills training group to review the skills learned during therapy. Homework will be assigned between sessions to review these new strategies and skills. Participants will meet regularly with a psychiatrist to receive fluoxetine, discuss any side effects, and adjust dosage if necessary.
* Group 2 participants will receive DBT and placebo medication.
* Group 3 participants will receive supportive therapy and fluoxetine. Supportive therapy is nondirective and focuses on strengths, coping abilities, and current areas of difficulty in life in an unstructured format. Participants in this group will meet with an individual therapist each week for 50 minutes. Patients will also be assigned to a psychiatrist to receive fluoxetine every other week.
* Group 4 participants will receive supportive psychotherapy and placebo medication.

All patients participating in this study will continue treatment for 12 months and will be evaluated bimonthly. After 12 months, participants will undergo neuropsychological testing to identify any changes that occurred over the last year. The clinical status of each participant will also be assessed at 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for diagnosis of borderline personality disorder
* History of at least one suicide attempt or self-mutilation episode 12 months prior to study entry
* Experiences continued urges to self-mutilate or attempt suicide
* Stable living situation
* Use of effective birth control if sexually active
* Clinically stable enough to tolerate placebo condition
* Not participating in other forms of treatment during the study

Exclusion Criteria:

* Any current organic mental syndromes, lifetime schizophrenic or bipolar disorders, psychotic disorders, or mental retardation
* Inability to complete psychiatric interview due to lack of cooperation or lack of comprehension
* Unable to tolerate fluoxetine or DBT
* Currently receiving treatment for an acute medical illness or other debilitating problem, including substance abuse or anorexia nervosa
* History of major depression lasting more than 3 months
* Current Hamilton depression score above 22 and not receiving treatment
* Pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2001-03; Primary Completion 2008-01 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Stanley, PhD, Principal Investigator — Research Foundation for Mental Hygiene/Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the emergency department, clinician referrals and advertisements. Recruitment period ended 6 months prior to study end date.
Pre-assignment Details: 91 participants signed consent, 86 were randomized, 11 participants dropped out prior to treatment start. Therefore 75 participants remained, accounting for the discrepancy between the original 91 participants and the final count of 75. Participants were washed out of all psychotropic medications. Benzodiazepine is permitted for sleep.
Groups:
- DBT Fluoxetine: Dialectal behavior therapy (DBT) is a form of Cognitive behavior therapy targeting suicidal and non-suicidal self injury in borderline personality disorder and is delivered over a 12 month period,and fluoxetine, an SSRI that is given in standard dosing 20, 40, 60, 80 mg for 12 months.
  Fluoxetine: Fluoxetine is administered in standard dosing 20, 40, 60, 80 mg increased monthly if tolerated
  Dialectical Behavior Therapy: Dialectical Behavior Therapy is a form of CBT originally developed to treat suicidal and self injuring individuals with borderline personality disorder. Treatment consists of 2 sessions/week: individual psychotherapy and skills training group.
- DBT Placebo: Dialectal behavior therapy and placebo Dialectal behavior therapy (DBT) is a form of Cognitive behavior therapy targeting suicidal and non-suicidal self injury in borderline personality disorder and is delivered over a 12 month period, and placebo for fluoxetine, an SSRI that is given in standard dosing 20, 40, 60, 80 mg for 12 months.
  Dialectical Behavior Therapy: Dialectical Behavior Therapy is a form of CBT originally developed to treat suicidal and self injuring individuals with borderline personality disorder. Treatment consists of 2 sessions/week: individual psychotherapy and skills training group.
Period: Overall Study
Arm/Group | DBT Fluoxetine | DBT Placebo | Supportive Therapy Fluoxetine | Supportive Therapy Placebo
Started | 18 | 19 | 20 | 18
Completed | 14 | 14 | 14 | 13
Not Completed | 4 | 5 | 6 | 5

BASELINE CHARACTERISTICS:
Population: Suicidal and/or self injuring individuals with borderline personality disorder.
Groups:
- Dialectical Behavior Therapy Fluoxetine: Dialectal behavior therapy (DBT) is a form of Cognitive behavior therapy targeting suicidal and non-suicidal self injury in borderline personality disorder and is delivered over a 12 month period,and fluoxetine, an SSRI that is given in standard dosing 20, 40, 60, 80 mg for 12 months.
  Fluoxetine: Fluoxetine is administered in standard dosing 20, 40, 60, 80 mg increased monthly if tolerated
  Dialectical Behavior Therapy: Dialectical Behavior Therapy is a form of CBT originally developed to treat suicidal and self injuring individuals with borderline personality disorder. Treatment consists of 2 sessions/week: individual psychotherapy and skills training group.
- Total: Total of all reporting groups
Arm/Group | Dialectical Behavior Therapy Fluoxetine | Dialectical Behavior Therapy Placebo | Supportive Therapy Fluoxetine | Supportive Therapy Placebo | Total
Number analyzed (Participants) | 18 | 19 | 20 | 18 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (6.9) | 29.1 (8.3) | 32.3 (8.6) | 31.8 (11.2) | 30.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 17 | 13 | 58
  Male | 3 | 6 | 3 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Suicide Attempts
Description: Suicide attempt count total over the course of the 12 month treatment period (sum of 6 bimonthly assessments during the treatment phase)
Time Frame: Assessed bimonthly
Population: Suicidal and/or self injuring individuals with borderline personality disorder.
Measure: Number; unit: suicide attempt
Groups:
- Dialectical Behavior Therapy With Fluoxetine: Participants received 12 months of DBT and Fluoxetine medication with weekly medication visits (medication condition double blind)
- Dialectical Behavior Therapy With Placebo: Participants received 12 months of DBT and placebo with weekly medication visits (medication condition double blind)
- Supportive Therapy With Fluoxetine: Participants received 12 months of ST with fluoxetine medication with weekly medication visits (medication condition double blind)
- Supportive Therapy With Placebo: Participants received 12 months of ST placebo medication with weekly medication visits (medication condition double blind)
Arm/Group | Dialectical Behavior Therapy With Fluoxetine | Dialectical Behavior Therapy With Placebo | Supportive Therapy With Fluoxetine | Supportive Therapy With Placebo
Number analyzed (Participants) | 18 | 19 | 20 | 18
suicide attempt | 2 | 1 | 4 | 1

ADVERSE EVENTS:
Time Frame: During study enrollment (12 months)
Groups:
- Dialectical Behavior Therapy With Fluoxetine: Participants received 12 months of DBT therapy with fluoxetine with weekly medication management sessions (double blind). Primary planned analyses were with supportive therapy/placebo. Also, the fluoxetine and placebo medication arms were collapsed into one in order to test the hypothesis regarding differences in the primary outcome variable between the two psychotherapy groups. Similarly the psychotherapy conditions were collapsed to compare fluoxetine vs. placebo, to test the hypothesis regarding differences in the primary outcome measure between the two medication groups.
- Supportive Therapy With Fluoxetine: Participants received 12 months of supportive therapy with fluoxetine weekly medication management sessions(double blind). Planned analyses were with supportive therapy/placebo. Also, fluoxetine and placebo medication arms were collapsed into one in order to test the hypothesis regarding differences in the primary outcome variable between the two psychotherapy groups. Similarly the psychotherapy conditions were collapsed to compare fluoxetine vs. placebo. to test the hypothesis regarding differences in the primary outcome measure between the two medication groups..
- Dialectical Behavior Therapy With Placebo: Participants received 12 months of DBT therapy with placebo medication with weekly medication management sessions (double blind). Also, the fluoxetine and placebo medication arms were collapsed into one in order to test the hypothesis regarding differences in the primary outcome variable between the two psychotherapy groups.Similarly the psychotherapy conditions were collapsed to compare fluoxetine vs. placebo, to test the hypothesis regarding differences in the primary outcome measure between the two medication groups.
- Supportive Therapy With Placebo: Participants received 12 months of supportive therapy with placebo weekly medication management sessions(double blind). This condition served as the control condition. Also, the fluoxetine and placebo medication arms were collapsed into one in order to test the hypothesis regarding differences in the primary outcome variable between the two psychotherapy groups.Similarly the psychotherapy conditions were collapsed to compare fluoxetine vs. placebo, to test the hypothesis regarding differences in the primary outcome measure between the two medication groups.
Arm/Group | Dialectical Behavior Therapy With Fluoxetine | Supportive Therapy With Fluoxetine | Dialectical Behavior Therapy With Placebo | Supportive Therapy With Placebo
Serious Adverse Events (participants affected / at risk) | 1/18 | 2/20 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/20 | 0/19 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dialectical Behavior Therapy With Fluoxetine (N=18) | Supportive Therapy With Fluoxetine (N=20) | Dialectical Behavior Therapy With Placebo (N=19) | Supportive Therapy With Placebo (N=18)
Hospitalization or ED visitn (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No